CLINICAL TRIAL: NCT04997616
Title: Determination of Cannabinoid and Cannabinoid Metabolite Levels in Healthy Volunteers
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Company withdrew interest in the study
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 261847
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Healthy
Keywords: Cannabidiol; Hemp-based

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 25 mg/day dose of Happy Lane CBD (Lower Dose) (Experimental): One 25 mg Happy Lane CBD gel capsule per day (25 mg/day total dose) for 10 consecutive days at approximately the same time of day (±1 hour) on each of these days.
  Interventions: Dietary Supplement: Happy Lane Hemp Extract/CBD soft gels (25 mg/capsule)
- 50 mg/day dose of Happy Lane CBD (Larger Dose) (Experimental): Two 25 mg Happy Lane CBD gel capsules per day (50 mg/day total dose) for 10 consecutive days at approximately the same time of day (±1 hour) on each of these days. Both capsules will be taken at the same time as each other.
  Interventions: Dietary Supplement: Happy Lane Hemp Extract/CBD soft gels (25 mg/capsule)

INTERVENTIONS:
Dietary Supplement: Happy Lane Hemp Extract/CBD soft gels (25 mg/capsule) — Half of the study participants (5 women and 5 men) will be taking one gel capsule per day (25 mg/day dose), while the other half (5 women and 5 men) will be taking 2 gel capsules per day (50 mg/day dose). Study participants will be taking gel capsules for 10 consecutive days. At the end of this 10-day regimen, study participant will return to the TRI where blood specimen (up to 15 mL) will be collected within 2 to 6 hours after the last dose. Major plant cannabinoids and cannabinoid metabolites in each blood specimen will be determined using liquid chromatography-mass spectrometry.

SUMMARY:
Levels of major cannabinoid and cannabinoid metabolites (i.e., CBD, CBD-OH) will be determined in the plasma of healthy volunteers following 10 days of Happy Lane Hemp Extract/CBD soft gels (25 mg per capsule) supplementation using liquid chromatography-mass spectrometry (LCMS).

DETAILED DESCRIPTION:
The objective of the study is to determine the levels of CBD, CBD-OH, THC, THC-COOH, and 11-OH-THC in plasma of healthy volunteers that have ingested hemp extract/CBD for 10 consecutive days.

The research team is planning to recruit 24 adults (12 females, 12 males), age of 18-45 years old, inclusive to allow for enrollment of 20 eligible adults (10 females, 10 males). Subjects will be identified and recruited using AR Research via the UAMS Translational Research Institute (TRI). Specifically, TRI coordinators will assist with calling, screening, and scheduling potential subjects based on the list generated from AR Research.

After signing the informed consent form, which includes an attestation that the subject has not used cannabinoids within the past 4 weeks and an attestation that the subject will not use any prescription or over-the-counter medications during the study, each subject will provide a baseline plasma sample (up to 15 mL, collected by TRI coordinators) that will be used to determine if any cannabinoids (CBD, CBD-OH, THC, THC-COOH, and 11-OH-THC) are present in the blood.

All blood samples (pre- and post-intervention) will be analyzed at the completion of the study. Therefore, if cannabinoids are found in any of the baseline samples, the result will be noted but will not necessarily result in any subjects being excluded from the study. However, exclusion of data from subjects whose initial test show a positive result for CBD or THC from the overall study may be deemed necessary by the research team under certain circumstances (e.g., if the baseline THC and/or CBD signal in a study subject is so large that accurate detection of the intervention would be hindered).

After the informed consent form is signed and the baseline plasma sample is drawn, each subject will be provided with Happy Lane™ Hemp Extract/CBD soft gels (25 mg CBD per capsule; the certificate of analyses is provided along with this Study Protocol). Half of the subjects (5 women and 5 men) will be taking one gel capsule per day (25 mg/day dose), while the other half (5 women and 5 men) will be taking 2 gel capsules per day (50 mg/day dose, both capsules will be taken at the same time). Group assignment will be made randomly based on a computer-generated randomization list.

Subjects will take gel capsules for 10 consecutive days at approximately the same time of day (±1 hour) on each of these days, beginning the morning after consent is provided (Day 2). During this 10-day period, subjects will record number of capsules (1 or 2) and time of day ingested, as well as any adverse event in a diary. This diary will be provided to each subject at the time of consent (Day 1), and each subject will return for a second visit within 2 to 6 hours after the last dose of the 10-day regimen (Day 11). During the second visit, subject will return to TRI, and a blood specimen (up to 15 mL) will be collected. Diaries, empty capsule bottles, and any extra/unused capsules will also be returned to the study staff during this second visit (Day 11), so that capsule count may be conducted by study staff for drug accountability. Subjects will receive a follow-up phone call (Day 13 or next business day) to collect any adverse events (AE) that occurred after diaries were returned.

The blood specimens will be used for determination of major cannabinoids using the liquid chromatography-mass spectrometry. The cannabinoid/metabolite analysis will be performed at a certified laboratory in Oxford, Mississippi - ElSohly Laboratories, Inc (http://www.elsohly.com/). This is a DEA licensed analytical laboratory under leadership of Dr. Mahmoud ElSohly.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females, between 18- and 45-years old, inclusive
* Ability to provide consent for oneself, including:

  * Attestation not to use other cannabinoid-containing product(s) throughout the duration of the study
  * Attestation not to use prescription or over the counter medication(s) and/or supplements throughout the duration of the study

Exclusion Criteria:

* Self-reported use of any cannabinoids (i.e., CBD, THC) within the last 4 weeks.
* Use of any prescription (or over the counter) medication or supplements during the study or in the 24 hours before enrollment in the study
* Serious illness (e.g., abnormal liver or kidney function, cardiovascular disease, diabetes, etc.)
* Any other condition that in the opinion of the investigator might interfere with the safe conduct of the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Amount of CBD in plasma of healthy volunteers that have ingested hemp extract/CBD for 10 consecutive days using LCMS | 13 days
  Half of the study participants (5 women and 5 men) will be taking one gel capsule per day (25 mg/day dose), while the other half (5 women and 5 men) will be taking 2 gel capsules per day (50 mg/day dose). At the end of this 10-day regimen, study participant will return to the TRI where blood specimen (up to 15 mL) will be collected within 2 to 6 hours after the last dose. LCMS will be used to measure the presence of CBD in the plasma samples.
Amount of CBD-OH in plasma of healthy volunteers that have ingested hemp extract/CBD for 10 consecutive days using LCMS | 13 days
  Half of the study participants (5 women and 5 men) will be taking one gel capsule per day (25 mg/day dose), while the other half (5 women and 5 men) will be taking 2 gel capsules per day (50 mg/day dose). At the end of this 10-day regimen, study participant will return to the TRI where blood specimen (up to 15 mL) will be collected within 2 to 6 hours after the last dose. LCMS will be used to measure the presence of CBD-OH in the plasma samples.
Amount of THC in plasma of healthy volunteers that have ingested hemp extract/CBD for 10 consecutive days using LCMS | 13 days
  Half of the study participants (5 women and 5 men) will be taking one gel capsule per day (25 mg/day dose), while the other half (5 women and 5 men) will be taking 2 gel capsules per day (50 mg/day dose). At the end of this 10-day regimen, study participant will return to the TRI where blood specimen (up to 15 mL) will be collected within 2 to 6 hours after the last dose. LCMS will be used to measure the presence of THC in the plasma samples.
Amount of THC-COOH in plasma of healthy volunteers that have ingested hemp extract/CBD for 10 consecutive days using LCMS | 13 days
  Half of the study participants (5 women and 5 men) will be taking one gel capsule per day (25 mg/day dose), while the other half (5 women and 5 men) will be taking 2 gel capsules per day (50 mg/day dose). At the end of this 10-day regimen, study participant will return to the TRI where blood specimen (up to 15 mL) will be collected within 2 to 6 hours after the last dose. LCMS will be used to measure the presence of THC-COOH in the plasma samples.
Amount of 11-OH-THC in plasma of healthy volunteers that have ingested hemp extract/CBD for 10 consecutive days using LCMS | 13 days
  Half of the study participants (5 women and 5 men) will be taking one gel capsule per day (25 mg/day dose), while the other half (5 women and 5 men) will be taking 2 gel capsules per day (50 mg/day dose). At the end of this 10-day regimen, study participant will return to the TRI where blood specimen (up to 15 mL) will be collected within 2 to 6 hours after the last dose. LCMS will be used to measure the presence of 11-OH-THC in the plasma samples.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Koturbash, MD, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No